CLINICAL TRIAL: NCT00709306
Title: The Skin Savvy Study: A Behavioral Skin Cancer Prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carolyn Heckman, Associate Professor, Fox Chase Cancer Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: K07CA108685 (NIH); K07CA108685 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Skin Cancer Prevention
MeSH Terms: interventions — Motivational Interviewing; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Education (Placebo Comparator): Participants were given a packet of standard skin cancer prevention educational brochures and handouts from major professional organizations to review independently for 10-15 minutes.
  Interventions: Behavioral: Education
- Motivational Interviewing (Active Comparator): Participants met with a trained counselor who reviewed any personalized feedback of risk derived from the baseline assessments (e.g., history of sunburns, self-reported UV exposure, protective behaviors). Counselors utilized the basic motivational interviewing skills of open-ended questions, reflection of participant statements, affirmations/positive feedback, and summation of major points throughout the discussion. These sessions took about 22 minutes.
  Interventions: Behavioral: Motivational Interviewing
- UV-detect photos (Active Comparator): Participants were shown a regular black and white photo and a black and white UV-filtered photo of their face. Participants were told that "Any dark, spotted, freckled, wrinkled, uneven, or pitted areas indicate existing underlying skin damage that is difficult to reverse. However, protecting the skin from UV radiation can prevent future damage." Participants were asked what they noticed about the photos, what their reactions were, and how this might affect their behavior. These sessions took 12 minutes on average.
  Interventions: Device: UV-Detect Photos
- UV-detect photos & MI (Experimental): Participants met with a trained counselor who reviewed any personalized feedback of risk derived from the baseline assessments (e.g., history of sunburns, self-reported UV exposure, protective behaviors). Counselors utilized the basic motivational interviewing skills of open-ended questions, reflection of participant statements, affirmations/positive feedback, and summation of major points throughout the discussion. In addition to baseline feedback, participants were also interviewed about the black & white and UV-filtered photos of their faces. These sessions took about 25 minutes.
  Interventions: Device: UV-Detect Photos; Behavioral: Motivational Interviewing

INTERVENTIONS:
Device: UV-Detect Photos — UV-Detect Photos
  Arms: UV-detect photos; UV-detect photos & MI
Behavioral: Motivational Interviewing — Motivational Interviewing
  Arms: Motivational Interviewing; UV-detect photos & MI
Behavioral: Education — Education
  Arms: Education

SUMMARY:
The purpose of the proposed project is to investigate the efficacy and longevity of two novel approaches to changing skin protection behaviors: 1) UV-detect photos that reveal currently existing skin damage and 2) motivational interviewing (MI), a person-centered, yet directive counseling style used to enhance internal motivation to change health behaviors. The proposed investigations include a pilot study to refine the methodology; a small formal randomized controlled efficacy trial; and a dismantling study. These studies will also expand current knowledge and research in several major ways: 1) the use of UV-detect photos will enable highly salient and personalized feedback, 2) MI will be used in a previously untried health domain (skin cancer prevention), 3) objective skin color changes will be measured using state-of-the-art skin reflectance spectrophotometry, and 4) the proposed studies will test aspects of several major psychological theories (e.g., Transtheoretical Model, Prototype/Willingness Model) to identify moderators/mediators of outcome.

DETAILED DESCRIPTION:
Teens and young adults are at high risk for overexposure to ultraviolet (UV) radiation, a leading factor in the development of skin cancer. The majority of these individuals continue to protect themselves minimally and tan intentionally, including significant increases in tanning booth use recently. Such care-free behaviors exist despite widespread education/awareness about UV radiation and skin cancer. The purpose of the proposed project is to investigate the efficacy and longevity of two novel approaches to changing skin protection behaviors: 1) UV-detect photos that reveal currently existing skin damage and 2) motivational interviewing (MI), a person-centered, yet directive counseling style used to enhance internal motivation to change health behaviors. The proposed investigations include a pilot study to refine the methodology; a small formal randomized controlled efficacy trial; and a dismantling study. These studies will also expand current knowledge and research in several major ways: 1) the use of UV-detect photos will enable highly salient and personalized feedback, 2) MI will be used in a previously untried health domain (skin cancer prevention), 3) objective skin color changes will be measured using state-of-the-art skin reflectance spectrophotometry, and 4) the proposed studies will test aspects of several major psychological theories (e.g., Transtheoretical Model, Prototype/Willingness Model) to identify moderators/mediators of outcome. Therefore, the studies should provide useful information about process and outcome for skin cancer prevention researchers and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older

Exclusion Criteria:

* Visual impairment

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Heckman, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were consented, baselined, and randomized upon arrival to the in-person session, thus no enrolled participants were excluded from the study before assignment to one of the four treatment conditions.
Groups:
- Education Control: Participants were given a packet of standard skin cancer prevention educational brochures and handouts from major professional organizations to review independently for 10-15 minutes.
- UV-detect Photos and Motivational Interviewing: Participants met with a trained counselor who reviewed any personalized feedback of risk derived from the baseline assessments (e.g., history of sunburns, self-reported UV exposure, protective behaviors). Counselors utilized the basic motivational interviewing skills of open-ended questions, reflection of participant statements, affirmations/positive feedback, and summation of major points throughout the discussion. In addition to baseline feedback, participants were also interviewed about the black & white and UV-filtered photos of their faces. These sessions took about 25 minutes.
Period: Overall Study
Arm/Group | Education Control | Motivational Interviewing | UV-detect Photos | UV-detect Photos and Motivational Interviewing
Started | 48 | 44 | 58 | 47
Completed | 39 | 30 | 48 | 37
Not Completed | 9 | 14 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Educational Control: Participants were given a packet of standard skin cancer prevention educational brochures and handouts from major professional organizations to review independently for 10-15 minutes.
- Total: Total of all reporting groups
Arm/Group | Educational Control | Motivational Interviewing | UV-detect Photos | UV-detect Photos and Motivational Interviewing | Total
Number analyzed (Participants) | 48 | 44 | 58 | 47 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 44 | 58 | 47 | 197
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.29 (1.68) | 20.32 (1.41) | 20.43 (1.49) | 20.85 (1.67) | 20.47 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 49 | 44 | 162
  Male | 14 | 9 | 9 | 3 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 4 | 0 | 3 | 2 | 9
  Asian-American/Pacific Islander | 8 | 6 | 5 | 5 | 24
  Caucasian/White | 31 | 32 | 44 | 39 | 146
  Hispanic/Latino | 1 | 0 | 2 | 0 | 3
  Other/Mixed | 4 | 6 | 4 | 1 | 15
Stage of Change Scale [Count of Participants; unit: Participants] — The Sun Stage of Change (SOC) Scale has 4 items asking participants whether they have been protecting their skin for the past year (maintenance), if they protect their skin now (action), whether they intend to protect their skin in the next 30 days (preparation), whether they intend to protect their skin in the next year (contemplation), or none of the above (pre-contemplation).
  Participants
    Precontemplation | 17 | 15 | 24 | 15 | 71
    Contemplation | 5 | 4 | 4 | 4 | 17
    Preparation | 8 | 12 | 14 | 14 | 48
    Action | 5 | 3 | 6 | 2 | 16
    Maintenance | 13 | 10 | 9 | 10 | 42
    data missing | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Sun Stage of Change at 3 Months
Description: The Sun Stage of Change (SOC) Scale has 4 items asking participants whether they have been protecting their skin for the past year (maintenance), if they protect their skin now (action), whether they intend to protect their skin in the next 30 days (preparation), whether they intend to protect their skin in the next year (contemplation), or none of the above (pre-contemplation).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Education Control | Motivational Interviewing | UV-detect Photos | UV-detect Photos and Motivational Interviewing
Number analyzed (Participants) | 44 | 38 | 50 | 43
Participants
  Precontemplation | 17 | 5 | 10 | 12
  Contemplation | 2 | 1 | 3 | 2
  Preparation | 7 | 15 | 15 | 15
  Action | 3 | 7 | 8 | 4
  Maintenance | 15 | 10 | 14 | 10

2. Primary Outcome: Sun Stage of Change at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Education Control | Motivational Interviewing | UV-detect Photos | UV-detect Photos and Motivational Interviewing
Number analyzed (Participants) | 39 | 30 | 48 | 37
Participants
  Precontemplation | 10 | 4 | 11 | 7
  Contemplation | 2 | 3 | 2 | 0
  Preparation | 7 | 5 | 11 | 20
  Action | 6 | 3 | 7 | 5
  Maintenance | 14 | 15 | 17 | 5

ADVERSE EVENTS:
Time Frame: Because this protocol involves low risk assessments and interventions (e.g., survey, brochure, UV picture, MI counseling, spectrophotometry), adverse event data were not collected. Because discussing cancer risk and looking at photos of UV damage may be upsetting, participants were monitored for distress at the time of baseline/intervention and any participants, however, no participants exhibited undue anxiety or concern during their participation.
Description: Because discussing cancer risk and looking at photos of UV damage may be upsetting, participants were monitored for distress at the time of baseline/intervention and any participants, however, no participants exhibited undue anxiety or concern during their participation.
Arm/Group | Education Control | Motivational Interviewing | UV-detect Photos | UV-detect Photos and Motivational Interviewing
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No